CLINICAL TRIAL: NCT06280430
Title: Serum Elafin :A Biomarker in Behcet Disease and Its Relation to Vascular Involvement and Disease Activity
Brief Title: Vascular Affection in Behcet Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lobna Amer Araby Ahmed, Assuit, Assiut University
Other Study IDs: Vascular affection in behcet
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Behcet Disease and Vascular Involvement
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with behcet disease
- Healthy control group

SUMMARY:
To measure the level of serum elafin in patients with behcet disease and to assess the correlation between serum elafin and vascular affection and their relation with disease activity

DETAILED DESCRIPTION:
Behcet disease is a chronic multi systemic inflammatory disease characterized by recurrent oral and genital ulcers and multiple systemic affection . Elafin is a serine protease inhibitor produced mainly by epithelial cells . previous studies documented the role of serum elafin in pathogenesis of behcet disease.vascular complications may be one if the earliest manifestation leading to the diagnosis of behcet disease.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as behcet disease Age (20-45)

Exclusion Criteria:

* age <20 and >45 Other autoimmune diseases Risk factors (ischemic heart disease, diabetes) Chronic conditions (malignancy, chronic kidney disease)

Ages: 20 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: 45 patients with behcet disease aged(20-45) in comparison with 45 heathy participant s
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
To measure the level of serum elafin in behcet patients and compare it with control group | Within 1year
  Measure the level of serum elafin in behcet and its relation to disease activity and vascular involvement